CLINICAL TRIAL: NCT02371408
Title: A Phase IIb/IIIa, Randomized Study to Evaluate the Efficacy and Safety of PPI-668 (NS5A Inhibitor) Plus Sofosbuvir, With or Without Ribavirin, in Patients With Chronic Hepatitis C Genotype-4
Brief Title: A Study of the Efficacy and Safety of PPI-668 (NS5A Inhibitor) Plus Sofosbuvir, With or Without Ribavirin, in Patients With Chronic Hepatitis C Genotype-4
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharco Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPI-668-202
Record Dates: First submitted 2015-02-01; First posted 2015-02-25 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ravidasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1a: Treatment-naive patients, without ribavirin (RBV) (Experimental): PPI-668 + sofosbuvir for 12 weeks
  Interventions: Drug: ravidasvir hydrochloride; Drug: sofosbuvir
- 1b: Treatment-naive patients, with RBV (Experimental): PPI-668 + sofosbuvir + ribavirin (RBV) for 12 weeks
  Interventions: Drug: ravidasvir hydrochloride; Drug: sofosbuvir; Drug: ribavirin
- 2a: Non-cirrhotic previous non-responders, without RBV (Experimental): PPI-668 + sofosbuvir for 12 weeks
  Interventions: Drug: ravidasvir hydrochloride; Drug: sofosbuvir
- 2b: Non-cirrhotic previous non-responders, with RBV (Experimental): PPI-668 + sofosbuvir + ribavirin for 12 weeks
  Interventions: Drug: ravidasvir hydrochloride; Drug: sofosbuvir; Drug: ribavirin
- 3a: Cirrhotic previous non-responders 12 weeks (Experimental): PPI-668 + sofosbuvir + ribavirin for 12 weeks
  Interventions: Drug: ravidasvir hydrochloride; Drug: sofosbuvir; Drug: ribavirin
- 3b: Cirrhotic previous non-responders 16 weeks (Experimental): PPI-668 + sofosbuvir + ribavirin for 16 weeks
  Interventions: Drug: ravidasvir hydrochloride; Drug: sofosbuvir; Drug: ribavirin

INTERVENTIONS:
Drug: ravidasvir hydrochloride — 200 mg
  Other Names: PPI-668
Drug: sofosbuvir — 400 mg
Drug: ribavirin — 1000 mg - 1200 mg per day, weight-based dosing
  Arms: 1b: Treatment-naive patients, with RBV; 2b: Non-cirrhotic previous non-responders, with RBV; 3a: Cirrhotic previous non-responders 12 weeks; 3b: Cirrhotic previous non-responders 16 weeks

SUMMARY:
The study will assess the efficacy of PPI-668 (USAN: ravidasvir hydrochloride) in combination with sofosbuvir, with or without ribavirin, in the following Egyptian HCV gt-4 patient populations:

1. Treatment-naïve patients, with and without cirrhosis (Group 1)
2. Previous non-responders to interferon-based therapies, without cirrhosis (Group 2)
3. Previous non-responders to interferon-based therapies, with cirrhosis (Group 3)

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 18 years & ≤ 65 years of age.
2. HCV antibody positive, with serum HCV RNA ≥ 10,000 IU/mL, with clinical history compatible with chronic hepatitis C.
3. HCV genotype-4 infection, confirmed at the central study laboratory
4. Body mass index (BMI) between 18 and 35 kg/m2, inclusive.
5. Both male and female patients who have childbearing potential must agree to practice an acceptable method of birth control during the study and for at least 6 months after the cessation of treatment; such contraceptive methods must include at least one barrier method.
6. Patients for Group 1 must be treatment-naïve - i.e., they have never received any antiviral treatment for their HCV infection, including interferon, pegylated interferon, ribavirin, or other regulatory-approved or investigational HCV antiviral therapies.
7. Patients for Groups 2 and 3 must have previously failed treatment with an interferon-based therapy - i.e., interferon or pegylated interferon, with or without ribavirin, with no other previous HCV antiviral therapies.

   Patients for Group 2 must be non-cirrhotic diagnosed on screening visit by both Fibroscan™ liver stiffness measurement < 12.5 kPa and FIB-4 score < 3.25 if the results of Fibroscan and FIB-4 score are not matching; liver biopsy will be used for detection of cirrhosis. In case that the liver biopsy is not applicable, hepatic imaging or ultrasound reports could be used for determination of cirrhosis.

   Patients for Group 3 must have underlying cirrhosis diagnosed on screening visit by both Fibroscan liver stiffness measurement > 12.5 kPa and FIB-4 score > 3.25, if the results of Fibroscan and FIB-4 score are not matching liver biopsy will be used for detection of cirrhosis. In case that the liver biopsy is not applicable, hepatic imaging or ultrasound reports could be used for determination of cirrhosis.
8. Willing and able to give informed consent
9. Willing and able to complete all study visits and procedures, including compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Mixed genotype or non-typable HCV genotype infection,
2. Positive test for HBsAg or HIV antibody, or IgM antibody to HAV or HEV
3. History of schistosomiasis or positive test for schistosoma surface antigen at Screen.
4. Serum alpha-fetoprotein (AFP) >100ng/ml. Patients with an AFP between 50 and 100ng/ml may be included as long as a liver ultrasound within 3 months of Screening, or at Screening, shows no evidence of potential hepatocellular cancer.
5. History of treatment with any investigational or regulatory-approved direct-acting antiviral (DAA) agent for HCV infection - nucleos(t)ide or non-nucleosidic HCV polymerase inhibitor, HCV protease inhibitor, NS5A inhibitor, or other antiviral agent for HCV infection other than pegylated -interferon and/or ribavirin Previous pegylated interferon and/or ribavirin treatment is allowed for Groups 2 and 3 but prohibited for group 1, as noted above in Inclusion criterion 6)
6. Evidence of a medical condition other than HCV that is contributing to liver disease
7. History of, or clinical signs of, hepatic decompensation or portal hypertension:

   Variceal bleeding, or documented esophageal or GI varices (at investigator discretion, patients suspected of having esophageal varices should be evaluated by endoscopy, and varices excluded) Ascites by history or on physical examination Documented or suspected hepatic encephalopathy

   Physical signs of portal hypertension:

   Clinically significant splenomegaly Spider angiomata History of porto-systemic shunt procedure(s)
8. Uncontrolled diabetes mellitus as evidenced by HgbA1C ≥ 8.5% at Screening.
9. Hemoglobin < 11g/dL for females and < 12 g/dL for males
10. WBC count < 3,500/mm3 OR absolute neutrophil count (ANC) < 1800/mm
11. Platelet count < 75,000/mm3
12. Serum creatinine > 1.3 x ULN OR creatinine clearance (GFR) < 50 mL/minute
13. Serum ALT or AST >10x ULN
14. Serum albumin ≤ 3.2 g/dl
15. Direct serum bilirubin > 2xULN
16. INR > 1.7.
17. History of poorly controlled asthma, with one or more hospitalizations or emergency room visits in the previous 6 months
18. History of any malignancy within the last 5 years (except prostate cancer still within Glisson's capsule or basal cell carcinoma of the skin).
19. History of alcohol abuse as assessed by the investigator within the past 2 years, or an alcohol use pattern that may interfere with the patient's study compliance. Patients must have abstained from alcohol for at least 6 months prior to study start.
20. History of drug abuse as assessed by the investigator within the last 2 years.
21. Pregnancy, including current lactation in female patients, male patients with partners who are pregnant, or female patients intending to become pregnant.
22. Major surgery requiring overnight hospitalization within 3 months prior to Screening
23. Participation in another clinical trial of an investigational drug or device within 6 months prior to Screening
24. Current use or history of use within the preceding 6 months of immunosuppressive or immune-modulating agents, including: azathioprine, systemic corticosteroids (prednisone or prednisone equivalent of more than 10mg/day for more than 10 days), or other immunosuppressive agents. Use of inhaled steroids for mild/moderate asthma and topical steroids for minor skin conditions is allowed.
25. History of solid organ or bone marrow transplantation.
26. History of use of medications associated with QT prolongation concurrently or within the 30 days prior to Screening Visit, including: macrolides, antiarrhythmic agents, azoles, fluoroquinolones, and tricyclic anti-depressants.
27. correction, or a personal or family history of Torsades de Pointe.
28. Cardiac ischemia with history of recurrent angina, clinically symptomatic cardiac abnormalities, or requirement for cardiac pacemaker
29. History of a known allergy to ribavirin (RBV), or any excipient in the investigational product, or history of drug or other allergy that, in the opinion of the investigator, mitigates against study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Proportions of patients who achieve Sustained Virologic Response at 12 weeks post-treatment (SVR12) | post-treatment week 12
  Sustained Virologic Response is defined as serum HCV RNA < LLOQ at post-treatment visits.

SECONDARY OUTCOMES:
Proportions of patients who achieve Sustained Virologic Response at 4 weeks post-treatment (SVR4) | post-treatment week 4
Proportions of patients who achieve Sustained Virologic Response at 24 weeks post-treatment (SVR 24) | post-treatment week 24
Proportion of treated study participants prematurely discontinuing study treatment for any reason, proportion prematurely discontinuing treatment for lack of efficacy or for clinical adverse events or laboratory abnormalities | during treatment and up to 24 weeks post-treatment
Proportion of patients experiencing treatment-emergent adverse events, and proportion of patients experiencing adverse events considered to be probably or possibly related to one or more of the study drugs | during treatment and up to 24 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, M.D., Principal Investigator — Kasr El Aini Viral Hepatitis Center
Locations (3):
- Egypt (3):
  - Al-Qahira Al-Fatimeya MoH Hospital, Cairo
  - Kasr El Aini Viral Hepatitis Center, Cairo
  - National Liver Institute, Menoufiya

REFERENCES:
- [Derived] Esmat G, Elbaz T, El Raziky M, Gomaa A, Abouelkhair M, Gamal El Deen H, Sabry A, Ashour M, Allam N, Abdel-Hamid M, Nada O, Helmy S, Abdel-Maguid H, Colonno R, Brown N, Ruby E, Vig P, Waked I. Effectiveness of ravidasvir plus sofosbuvir in interferon-naive and treated patients with chronic hepatitis C genotype-4. J Hepatol. 2017 Sep 19:S0168-8278(17)32286-9. doi: 10.1016/j.jhep.2017.09.006. Online ahead of print. PMID 28935432